CLINICAL TRIAL: NCT03604185
Title: Effects of Short-term Choir Participation on Auditory Perception in Hearing-aided Older Adults.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 forced the shut down of the study
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Sonova AG (Industry); Mitacs (Industry)
Responsible Party: Principal Investigator, Frank Russo, Doctor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAC 2018-089
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss; Auditory Perception; Music Therapy; Aging
Keywords: Hearing Loss; Auditory Processing; Aging; Speech Perception in Noise (SIN); Pitch Discrimination; Frequency Following Response (FFR); Choir Singing; Musical Training
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Sixty hearing aided older adults will be randomly assigned to one of three conditions: a choir singing class (n=20), a music appreciation class (n=20), and a do-nothing control group (n=20). Choir participants will take part in a singing class for 14 weeks, during which they will take part in group singing (2 hours/week) supported by individual online musical training (1 hour/week). Participants will undergo pre- and post-training assessments, conducted during the first week of the choir class and again after the last week. The music appreciation group will consist of hearing aided older adults attending 14 weeks of music listening classes, and the do-nothing control group will not be engaged in an active intervention. All participants will undergo the same battery of assessments, measured before and after the 14-week time frame.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Choir Singing Group (Experimental): Choir participants will take part in weekly two-hour group choral sessions over the course of fourteen weeks, during which time they will receive pitch training and vocal direction. In addition to the weekly group choir sessions, participants will be offered optional individual online musical and vocal training exercises (up to one hour weekly).
  Interventions: Behavioral: Choir Singing
- Music Appreciation Group (Active Comparator): Participants assigned to the music appreciation class will take part in a fourteen week course which will emphasize analytic listening to musical excerpts, which will match the choir class in terms of duration, homework demands, and instructor - both classes will be taught by the same person.
  Interventions: Behavioral: Music Appreciation
- Do-Nothing Control Group (No Intervention): The do-nothing control group will not receive any active training.

INTERVENTIONS:
Behavioral: Choir Singing — A weekly 2-hour group choral session over fourteen weeks. Plus an optional weekly 1-hour online musical and vocal training session.
  Arms: Choir Singing Group
Behavioral: Music Appreciation — A fourteen week course which will emphasize analytic listening to musical excerpts, and will match the choir class in terms of duration, homework demands, and instructor.
  Arms: Music Appreciation Group

SUMMARY:
Hearing loss has been associated with decreased emotional wellbeing and reduced quality of life in aging adults. Although hearing aids can target aspects of peripheral hearing loss, persistent perceptual deficits are widely reported. One prevalent example is the loss of the ability to perceive speech in a noisy environment, which severely impacts quality of life and goes relatively unremediated by hearing aids. Musicianship has been shown to improve aspects of auditory processing, but has not been studied as a short-term intervention for improving these abilities in older adults with hearing aids. The current study investigates whether short-term choir participation can improve three aspects of auditory processing: perception of speech in noise, pitch discrimination, and the neural response to brief auditory stimuli (frequency following response; FFR). Sixty hearing aided older adults (aged 50+) recruited from the Greater Toronto Area will be randomly assigned to one of three conditions: a choir singing class (n=20), a music appreciation class (n=20), and a do-nothing control group (n=20). Choir participants will take part in a singing class for 14 weeks, during which they will take part in group singing (2 hours/week) supported by individual online musical training (1 hour/week). Participants will undergo pre- and post-training assessments, conducted during the first week of the choir class and again after the last week. Participants in the music appreciation class will be involved in 14 weeks of music listening classes, and the do-nothing control group will not engaged in an active intervention. All participants will undergo the same battery of assessments, measured before and after the 14-week time frame. Auditory assessments (speech perception in noise and pitch discrimination tests) will be administered electronically, and the FFR will be obtained using electroencephalography (EEG). Each of the four assessment sessions (two pre-training, two post-training) will last approximately 1.5 hours, for a total of 6 hours of data collection. The goal of this research is to investigate whether short-term musical training will result in improved auditory outcomes for older adults with hearing aids. It is predicted that the choir singing group will demonstrate the greatest improvements across all auditory measures, and that both the choir singing and musical appreciation groups will experience greater improvements than the do-nothing control group.

DETAILED DESCRIPTION:
The study will investigate whether choir participation and musical training can improve three aspects of auditory processing in hearing aided older adults: perception of speech in noise, pitch discrimination, and the neural response to brief auditory stimuli (frequency following response; FFR). Sixty older adults with hearing aids will be recruited from the Greater Toronto Area through flyers in Connect Hearing Clinics and Ryerson's 50+ Program Bulletin, as well as through an ad in the Toronto Star, which will provide contact information for the Science of Music, Auditory Research and Technology (SMART) Laboratory. Anyone who contacts the SMART Lab with an interest in participating will be administered a pre-screening questionnaire over the phone by a study researcher; this may also be administered by email depending on participant preference. Those who are eligible and give informed consent will be randomly assigned to one of three groups: a choir singing class (n=20), a music appreciation class (n=20), or a do-nothing control condition (n=20). Each choir participant will come into the SMART Laboratory for two pre-training assessments that will take approximately 1.5 hours each, during which time they will complete several questionnaires and assessments of auditory abilities (including pitch discrimination and speech perception in noise), and undergo an electroencephalograph (EEG) during presentation of repeated auditory stimuli (obtaining the FFR). Choir participants will then take part in weekly two-hour group choral sessions over the course of fourteen weeks, during which time they will receive pitch training and vocal direction in an open and encouraging environment. In addition to the weekly group choir sessions, participants will be offered optional individual online musical and vocal training exercises (up to one hour weekly), designed to target and improve the participants' abilities to perceive and produce small changes in pitch. After fourteen weeks of choir participation and musical training, each choir participant will return to the SMART Lab for two post-training assessments that will last approximately 1.5 hours each. During post-training data collection sessions, participants will complete different versions of the pre-training auditory assessments, and undergo a post-training EEG. Participants assigned to the music appreciation class will take part in a fourteen week course which will emphasize analytic listening to musical excerpts, which will match the choir class in terms of duration, homework demands, and instructor - both classes will be taught by the same person. The do-nothing control group will undergo the same battery of pre- and post-testing, with fourteen weeks between data collection sessions, but will not receive any active training during this time. All participants in the music appreciation class and the do-nothing control group will be offered the opportunity to take part in the choir at a later date. It is hypothesized that musical training - in particular, group singing practice - will result in improved outcomes of auditory perceptual measures in hearing-aided older adults. It is predicted that individuals who take part in 14 weeks of group choral singing will demonstrate improvements across all auditory measures, including improved pitch discrimination, enhanced ability to perceive speech in noisy environments, and higher fidelity and more consistent neural responses to brief auditory stimuli (as indexed by features of the FFR). It is predicted that participants in the music appreciation class may demonstrate auditory improvements as a result of their focus on music perception, but that these improvements will not be as significant as those of the choir participants. It is further predicted that both training groups will outperform the do-nothing control group on post-training measures.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (50+)
* Have a hearing aid
* Hearing loss must be mild-moderate (i.e. between 25 and 60 dB HL at standard test frequencies)
* Hearing loss must be symmetrical (i.e. no more than 25 dB HL difference between ears at any standard test frequency)

Exclusion Criteria:

* Adults younger than 50
* Do not have a hearing aid
* Hearing loss exceeds mild-moderate rating (i.e. any standard test frequency measures higher than 25 - 60 dB HL)
* Hearing loss is asymmetrical (i.e. at any standard test frequency the difference between ears is larger than 25 dB HL).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Speech-in-noise perception: Signal-to-Noise Ratio (SNR) | 14 weeks
  Ability to track speech in a noisy environment will be assessed using the QuickSIN test (Speech-In-Noise; Etymotic Research; Killion, Niquette, Gudmundsen, Revit, & Banerjee, 2004) and the Revised Speech Perception in Noise (R-SPIN) test (Bilger, 1984).

SECONDARY OUTCOMES:
Pitch discrimination: Frequency Difference Limens (FDL) | 14 weeks
  Participants' ability to distinguish different frequencies will be measured using a computerized assessment of frequency difference limens (FDL).
Frequency Following Response (FFR) | 14 weeks
  The frequency following response (FFR) is a component of the auditory brainstem response, which represents the capacity of neurons in the auditory brainstem to track and encode changes in frequency during the solid state of a complex auditory signal (Skoe and Kraus, 2010). This is measured by obtaining an EEG during repeated presentation of brief complex auditory stimuli, and analyzing the signal for fidelity (as indexed by the FFT, a fast Fourier transform of the signal) and consistency (as indexed by the ITPC, inter-trial phase coherence).

CONTACTS AND LOCATIONS:
Overall Officials: Frank Russo, PhD, Principal Investigator — Toronto Metropolitan University; Ella Dubinsky, MA, Study Director — Toronto Metropolitan University
Locations (1):
- Toronto Metropolitan University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Killion MC, Niquette PA, Gudmundsen GI, Revit LJ, Banerjee S. Development of a quick speech-in-noise test for measuring signal-to-noise ratio loss in normal-hearing and hearing-impaired listeners. J Acoust Soc Am. 2004 Oct;116(4 Pt 1):2395-405. doi: 10.1121/1.1784440. PMID 15532670
- [Background] Bilger RC. (1984b) Speech recognition test development. In: Elkins E, ed. Speech Recognition by the Hearing Impaired. ASHA Reports 14. Rockville, MD: American Speech-Language-Hearing Association.
- [Background] Skoe E, Kraus N. Auditory brain stem response to complex sounds: a tutorial. Ear Hear. 2010 Jun;31(3):302-24. doi: 10.1097/AUD.0b013e3181cdb272. PMID 20084007